CLINICAL TRIAL: NCT06586801
Title: A Multicenter Prospective Cohort Study of the Patient-Reported Outcomes in ALK Positive Advanced Non-Small Cell Lung Cancer (NSCLC) in China
Brief Title: The Patient-Reported Outcomes in ALK Positive Advanced NSCLC in China
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ML44840
Record Dates: First submitted 2024-08-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ALK+ NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort I: 400 ALK-positive locally advanced or metastatic NSCLC patients who are treated with Alectinib
  Interventions: Other: Patient-reported outcome
- Cohort II: 200 ALK-positive locally advanced or metastatic NSCLC patients who are treated with Lorlatinib
  Interventions: Other: Patient-reported outcome
- Cohort III: 200 ALK-positive locally advanced or metastatic NSCLC patients who are treated with other ALK-TKIs except for Alectinib and Lorlatinib
  Interventions: Other: Patient-reported outcome

INTERVENTIONS:
Other: Patient-reported outcome — Patient-reported outcome data will be collected using the following instruments:EORTC QLQ-C30, EORTC QLQ-LC13, selected items from the PRO-CTCAE, EORTC-IL46.
  The first collection of the information in questionnaires (EORTC QLQ-C30, EORTC QLQ-LC13, PRO-CTCAE [select items]), which defined as baseline- PROs, will be completed at Cycle 1, Day 1±7days prior to administration of study drug; then the rest times of collection will be completed at every two treatment cycle prior to administration of study drug (i.e., on Cycle 3, Day 1±7days; Cycle 5, Day 1±7days; Cycle 7, Day 1±7days; Cycle 9, Day 1±7days; Cycle 11, Day 1±7days; Cycle 13, Day 1±7days) . EORTC-IL46 will be completed at Cycle 3, Day 1±7days (baseline) prior to administration of study drug; then at every other study treatment cycle prior to administration of study drug (i.e., on Cycle 5, Day 1±7days; Cycle 7, Day 1±7days; Cycle 9, Day 1±7days; Cycle 11, Day 1±7days; Cycle 13, Day 1±7days)

SUMMARY:
This is a multicenter, prospective, longitudinal observational study designed to evaluate the patient-reported outcomes and safety profiles of patients with ALK positive advanced Non-Small Cell Lung Cancer (NSCLC) who received ALK-TKIs as first-line treatment.

Approximately 800 patients with ALK-positive locally advanced or metastatic NSCLC will be enrolled in this study. This study has 3 parallel cohorts which are listed below.

Patient-reported outcome data will be collected using the following instruments: EORTC QLQ-C30, EORTC QLQ-LC13, selected items from the PRO-CTCAE, EORTC-IL46.

DETAILED DESCRIPTION:
A total of 800 patients with ALK+ NSCLC will be enrolled in this study. The actual number of sites can be increased or decreased as appropriate. In order to approach the real world medication situation, the number of patients treated with Alectinib will be 400 cases; the number of patients treated with Lorlatinib will be 200 cases; the number of patients treated with the other ALK-TKIs will be 200 cases in total.

Study Population The study population is intended to follow the real-world use of ALK-TKIs treatment; therefore, minimal inclusion and exclusion criteria will be used. The study population will comprise patients treated with ALK-TKIs for ALK-positive advanced NSCLC.

Patients in all 3 cohorts who meet any of the following criteria will be excluded from study entry:

* Patients receiving ALK-TKIs as investigational study drugs in a clinical trial for the treatment of advanced NSCLC
* Patients participating in clinical trials within 28 days prior to initiation of study treatment
* Pregnant, lactating, or breastfeeding women Statistical Methods Primary Analysis The primary objective for this study is to describe the patient-reported outcomes in patients with ALK+ locally advanced or metastatic NSCLC who received ALK-TKIs as first-line treatment in the real world situation. Analyses were conducted using the full analysis set (FAS), which comprised all 3 cohorts of patients enrolled in the study population with at least baseline data in eCRFs. The PRO analysis set consists of all patients in the FAS who completed at least one baseline questionnaire and at least one post baseline questionnaire.Patients with no post-baseline information will be censored at the date of enrollment.

Proportion of patients reporting clinically meaningful deterioration (decrease from baseline of ≥ 10 points) in the subscales of EORTC QLQ-LC13 (fatigue, chest pain) and QLQ-C30 (cognitive, physical and role functioning) will be summarized.

Change(s) from baseline scores will be conducted for fatigue, chest pain as measured by the EORTC QLQ-LC13 and cognitive functioning, physical and role functioning by QLQ-C30 at each assessment time point.

Presence, frequency of occurrence, severity, and/or degree of interference with daily function of symptomatic treatment toxicities (swelling, rash, blurred vision, anxious, sad) as assessed through use of the NCI PRO-CTCAE Frequency of patients' response of the degree they are troubled with treatment symptoms, as assessed through use of the single-item EORTC Item List (IL46) Summary statistics (number of patients, mean, standard deviation, median, minimum, maximum, 95% CI) will be applied for baseline characteristics and absolute score(s).

Secondary analysis Incidence and severity of adverse events based on the NCI CTCAE v5.0 and the rate of ALK-TKIs treatment changes by different reasons will be summarized to evaluate the safety and tolerability of ALK-TKIs as first-line treatment in each three cohorts. All variables will be summarized by number of patients, mean, standard deviation, median, minimum, maximum.

Analyses were conducted using SAS statistical software, version 9.4 (SAS Institute Inc, Cary, North Carolina).

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form (ICF) as per local regulations
* Female or male aged 18 years or older
* Ability to comply with the study protocol, in the judgment of the investigator
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0, 1, or 2
* Have a confirmed diagnosis of locally advanced or metastatic NSCLC on or after the date of local approval for ALK-TKIs as first-line monotherapy regimen for ALK-positive advanced NSCLC and planned to receive treatment as per routine for at least one cycle (28 days) while on study
* ALK positive as determined by Ventana immunohistochemistry (IHC), fluorescent in situ hybridization (FISH), reverse transcription polymerase chain reaction(RT-PCR) and next generation sequencing (NGS), documented prior to receiving treatment with an ALK inhibitor
* Planned to receive, treatment for ALK-positive advanced NSCLC with ALK-TKIs
* Able to be followed up at the participating site
* Patients with advanced NSCLC who have asymptomatic central nervous system (CNS) metastases are eligible for inclusion

Exclusion Criteria:

* Patients receiving ALK-TKIs as investigational study drugs in a clinical trial for the treatment of advanced NSCLC
* Patients participating in clinical trials within 28 days prior to initiation of study treatment
* Pregnant, lactating, or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients with ALK-positive advanced NSCLC who are treated with ALK-TKIs according to standard of care and in line with local product information.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-LC13 | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  Proportion of patients reporting clinically meaningful deterioration (decrease from baseline of ≥10 points) in the subscales of EORTC QLQ-LC13 (fatigue, chest pain) ;Change from baseline score (by 2 cycles) in the subscales of EORTC QLQ-LC13 (fatigue, chest pain) .
EORTC QLQ-C30 | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  Proportion of patients reporting clinically meaningful deterioration (decrease from baseline of ≥ 10 points) in the subscales of QLQ-C30 (cognitive, physical and role functioning);Change from baseline score (by 2 cycles) in the subscales of QLQ-C30 (cognitive, physical and role functioning).
NCI PRO-CTCAE | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  Presence, frequency of occurrence, severity, and/or degree of interference with daily function of symptomatic treatment toxicities (swelling, rash, blurred vision, anxious, sad) as assessed through use of the NCI PRO-CTCAE.
EORTC Item List (IL46) | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  Frequency of patients' response of the degree they are troubled with treatment symptoms, as assessed through use of the Protocol ML44840, Version 2.0 single-item EORTC Item List (IL46)

SECONDARY OUTCOMES:
To evaluate the safety of ALK-TKIs as first-line treatment in advanced ALK+ NSCLC | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  Incidence and severity of adverse events, based on the NCI CTCAE v5.0.
To evaluate the tolerability of ALK-TKIs as first-line treatment in advanced ALK+ NSCLC | The data collection period for an individual patient was approximately 12 months, which could be truncated by treatment switching, patient withdrawal from the study, or death.
  ALK-TKIs treatment changes (dose modifications and/or discontinuation of treatment) and the rationale for treatment changes.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital

IPD SHARING:
Plan to Share IPD: No